CLINICAL TRIAL: NCT00372086
Title: The Addition of Rosiglitazone to Insulin in Adolescents With Type 1 Diabetes and Poor Glycaemic Control: a Randomized, Placebo Controlled Trial
Brief Title: Rosiglitazone and Insulin in T1DM Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Collaborators: Sydney Children's Hospitals Network (Other); National Health and Medical Research Council, Australia (Other); Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 02/315; JHH ethics: 04/02/11/3.04; CHW ethics: 2003/037
Record Dates: First submitted 2006-09-03; First posted 2006-09-06 (Estimated); Last update posted 2006-09-06 (Estimated); Status verified 2006-09

CONDITIONS: Type 1 Diabetes; Puberty: >Tanner 2 Breast Development or Testis >4ml
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone

SUMMARY:
Type 1 Diabetes is the most common life-long disorder with onset in childhood. Patients need insulin injections, blood sugar monitoring several times each day, and adhere to a strict diet. Adequate control of blood glucose is essential to prevent long term kidney and eye complications that result in kidney failure and blindness. Adolescence is a time when diabetes is difficult to control, due in part to high growth hormone levels causing insulin resistance ( a state where the body does not respond as strongly to insulin). This study will test whether treatment with rosiglitazone (an oral medication used frequently in type 2 diabetes) will reduce the insulin resistance of adolescence and improve the control of type 1 diabetes during puberty.

ELIGIBILITY:
Inclusion Criteria:

* T1DM duration > 1year
* age 10-18years
* HbA1c > 8%
* puberty > Tanner stage 2 breast or testis >4ml

Exclusion Criteria:

* known non-compliance
* hypo unaware

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Enrollment: 32
Dates: Start 2003-08; Study Completion 2005-09

PRIMARY OUTCOMES:
HbA1c

SECONDARY OUTCOMES:
insulin dose
frequency of severe hypoglycaemia
insulin sensitivity assessed by euglycaemic, hyperinsulinaemic clamp
weight
BMI-SDS
skin fold thickness
cholesterol
adiponectin

CONTACTS AND LOCATIONS:
Overall Officials: Monique Stone, MBBS FRACP, Principal Investigator — Royal North Shore Hospital
Locations (1):
- Sydney Children's Hospital, Sydney, New South Wales, Australia